CLINICAL TRIAL: NCT02881775
Title: Immediate Effects of rTMS on Corticospinal Excitability of the Quadriceps in People With Knee Osteoarthritis
Brief Title: Immediate Effects of rTMS on Excitability of the Quadriceps With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16-0255
Record Dates: First submitted 2016-08-15; First posted 2016-08-29 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis, Knee
Keywords: TMS; rTMS; corticospinal; quadriceps
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Transcranial Magnetic Stimulation; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rTMS and exercise, then Sham rTMS and exercise (Experimental): At lab visit, subjects receive repetitive transcranial magnetic stimulation (rTMS) at 10 Hz, 5 sec on, 55 sec off and quadriceps isometric exercise (5% MVIC) for 15 minutes. This is followed by a wash out period of 1 week. At the next lab visit, subjects receive sham rTMS and exercise using the same parameters.
  Interventions: Device: rTMS and exercise; Device: Sham rTMS and exercise
- Sham rTMS and exercise, then rTMS and exercise (Sham Comparator): At lab visit, subjects receive sham repetitive transcranial magnetic stimulation (rTMS) at 10 Hz, 5 sec on, 55 sec off and quadriceps isometric exercise (5% MVIC) for 15 minutes. This is followed by a wash out period of 1 week. At the next lab visit, subjects receive the "true" rTMS and exercise using the same parameters.
  Interventions: Device: rTMS and exercise; Device: Sham rTMS and exercise

INTERVENTIONS:
Device: rTMS and exercise — rTMS at 10 Hz (5 sec on, 55 sec off) and light quadriceps isometric exercise (5% MVIC)
  Other Names: repetitive TMS
Device: Sham rTMS and exercise — rTMS unit is on and running but mu metal is placed between the coil and the skull
  Other Names: sham repetitive TMS

SUMMARY:
The purpose of the study is to identify things that influence the ability to "turn on" the thigh muscle (quadriceps). The thigh muscle tends to be under active with knee osteoarthritis, which may make it difficult to strengthen the muscle. The investigators are also testing a new technology called repetitive transcranial magnetic stimulation (rTMS) to determine whether it may help "turn up" activity in the under active thigh muscle immediately after its application. rTMS uses a targeted pulsed magnetic field, similar to what is used in an MRI (magnetic resonance imaging) machine to send an electrical signal from the brain to the thigh muscle.

DETAILED DESCRIPTION:
The investigators will recruit up to 20 people with symptomatic knee osteoarthritis. The 20 eligible participants will attend 3 sessions in the laboratory. Session 1 is to collect data for Aim 1. Sessions 2 and 3 will include the rTMS interventions and data collection for Aim 2.

Aim 1 is a descriptive study to compare the neural (cortical and corticospinal) excitability of the quadriceps in the symptomatic knee to the asymptomatic knee in participants with knee osteoarthritis. The investigators will examine the associations between neural excitability and clinical measures of pain, strength, function, and coping styles.

Aim 2 is a double blind, crossover study design. Each participant will partake in two testing sessions, spaced 1 week apart. The investigators will evaluate outcome measures prior to and following the "true" intervention versus the "sham" intervention. The true intervention is rTMS + exercise. The sham is sham rTMS + exercise. The primary outcome measures are quadriceps strength, as measured from a maximal isometric voluntary contraction, and quadriceps central activation ratio (CAR), as calculated from the torque values from the voluntary strength measurement and a brief, intense electrical stimulus. Secondary measures evaluate effects of the intervention on 1) clinical measures of pain and functional performance, 2) corticospinal excitability, and 3) intracortical inhibition and facilitation.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic knee osteoarthritis primarily involving one leg based on Western Ontario and McMaster Universities Arthritis Index (WOMAC) function subscale score > 10 (out of 100 points, indicating most dysfunction)
* diagnosis of knee osteoarthritis
* opposite knee with WOMAC pain score ≤ 5.
* opposite knee does not have a diagnosis of knee osteoarthritis

Exclusion Criteria:

* conditions affecting the leg other than osteoarthritis
* low blood pressure (< 90 systolic, 60 diastolic) or heart rate (< 60 beats per minute)
* conditions that limit exercise tolerance such as a heart condition
* pregnant or planning to become pregnant in the next 3 months
* conditions that alter sensation and pain processing
* BMI > 35
* severe arthritis in both knees
* history of leg or back surgery in the past year or knee replacement surgery;
* injection in the knee joint in the past 4 weeks
* requires an assistive device to walk
* any contraindications for TMS or rTMS (seizures, metal implants in head, brain related conditions, brain injury, drug or alcohol withdrawal)
* medications that lower seizure threshold
* history of fainting spells (syncope) or low blood pressure
* sleep deprived
* inability to understand and repeat back directions regarding the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L Givens, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | rTMS and Exercise, Then Sham rTMS and Exercise | Sham rTMS and Exercise, Then rTMS and Exercise
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0
Period: First Intervention (1-hr Session)
Arm/Group | rTMS and Exercise, Then Sham rTMS and Exercise | Sham rTMS and Exercise, Then rTMS and Exercise
Started | 9 (Two participants dropped out prior to First Intervention (1-hr Session).) | 7 (Two participants dropped out prior to First Intervention (1-hr Session).)
Completed | 9 | 7
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | rTMS and Exercise, Then Sham rTMS and Exercise | Sham rTMS and Exercise, Then rTMS and Exercise
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0
Period: Second Intervention (1-Hour Session)
Arm/Group | rTMS and Exercise, Then Sham rTMS and Exercise | Sham rTMS and Exercise, Then rTMS and Exercise
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants in the baseline population are the same as those in the intervention. All participants came for 3 laboratory sessions. The purpose of the first session was to collect baseline data on both the involved and uninvolved knee.
Groups:
- All Study Participants: Participants who were randomized to receive either rTMS and exercise or sham rTMS and exercise.
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] — intake questionnaire
  years | 63 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Quadriceps Central Activation Ratio (CAR)
Description: Quadriceps Central Activation Ratio (CAR) is a percentage of the amount of torque produced during the superimposed burst technique using maximal voluntary isometric contraction (MVIC) and superimposed burst torque. It is reported on a scale of 0 (worst) to 100% (best) activation.
Time Frame: Within 1 hour post intervention
Population: 4 subjects withdrew from the study after the baseline measures. This left 16 subjects for the intervention arm of the study. Four subjects declined to perform the test after the experience with the electrical stimulus in the baseline session.
Measure: Least Squares Mean (Standard Error); unit: % activation
Groups:
- rTMS and Exercise: At lab visit, subjects receive repetitive transcranial magnetic stimulation (rTMS) at 10 Hz, 5 sec on, 55 sec off and quadriceps isometric exercise (5% MVIC) for 15 minutes. This is followed by a wash out period of 1 week. At the next lab visit, subjects receive sham rTMS and exercise using the same parameters.
- Sham rTMS and Exercise: At lab visit, subjects receive sham repetitive transcranial magnetic stimulation (rTMS) at 10 Hz, 5 sec on, 55 sec off and quadriceps isometric exercise (5% MVIC) for 15 minutes. This is followed by a wash out period of 1 week. At the next lab visit, subjects receive the "true" rTMS and exercise using the same parameters.
Arm/Group | rTMS and Exercise | Sham rTMS and Exercise
Number analyzed (Participants) | 12 | 12
% activation
  CAR Baseline (BL) | 86.3554 (3.2921) | 86.1983 (3.2921)
  CAR BL Change | -1.2496 (2.1397) | -1.2670 (2.1397)
Statistical Analysis 1: Comparison: rTMS and Exercise vs Sham rTMS and Exercise; Comparison of CAR BL Change (treatment by time); Test type: Superiority; p = .9994, ANOVA — The threshold for significance was P <.05; Repeated measures ANOVA with restricted maximum likelihood estimation and Kenward-Roger standard errors. Degrees of freedom (DF) = 34.1

2. Primary Outcome: Quadriceps Maximal Voluntary Isometric Contraction (MVIC)
Description: HUMAC NORM electromechanical dynamometer is used to measure isometric torque generation in quadriceps muscle stabilized with 70 degrees of knee flexion. Units of measure are in Newton meters (Nm).
Time Frame: Within 1 hour post intervention
Population: 4 subjects withdrew from the study after the baseline measures. This left 16 subjects for the intervention arm of the study.
Measure: Least Squares Mean (Standard Error); unit: Nm
Arm/Group | rTMS and Exercise | Sham rTMS and Exercise
Number analyzed (Participants) | 16 | 16
Nm
  MVIC Baseline | 129.46 (11.8464) | 129.09 (11.8464)
  MVIC BL Change | -6.3473 (4.4266) | -6.1643 (4.4266)
Statistical Analysis 1: Comparison: rTMS and Exercise vs Sham rTMS and Exercise; Comparison of MVIC BL Change (treatment by time); Test type: Superiority; p = .9768, ANOVA — The threshold for statistical significance was p < .05; Repeated measures ANOVA with restricted maximum likelihood estimation and Kenward-Roger standard errors. DF = 45

3. Secondary Outcome: Numeric Pain Rating Scale (NPRS) Score
Description: Pain intensity is rated on a visual analog scale of 0-10 where 0 is no pain and 10 is maximum pain
Time Frame: Within 1 hour post intervention
Population: 4 subjects withdrew from the study after the baseline measures. This left 16 subjects for the intervention arm of the study. For two subjects, the research assistant missed obtaining the post-intervention pain rating.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | rTMS and Exercise | Sham rTMS and Exercise
Number analyzed (Participants) | 16 | 14
score on scale
  NPRS Baseline | 3.25 (.5749) | 3.000 (.5749)
  NPRS BL Change | -.625 (.4187) | -.1570 (.4378)
Statistical Analysis 1: Comparison: rTMS and Exercise vs Sham rTMS and Exercise; Comparison of NPRS BL Change (treatment by time); Test type: Superiority; p = 0.4440, ANOVA — threshold for statistical significance is p < .05; Repeated measures ANOVA with restricted maximum likelihood estimation and Kenward-Roger standard errors. DF = 43.1

4. Secondary Outcome: Pressure Pain Threshold (PPT) - Medial Knee
Description: Using the AlgoMed algometer, pressure at a rate of 35 kPA/second is applied to the medial knee to the level that subject indicates is painful. Units of measure are kilopascal (kPa)
Time Frame: Within 1 hour post intervention
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kPa
Arm/Group | rTMS and Exercise | Sham rTMS and Exercise
Number analyzed (Participants) | 16 | 16
kPa
  PPT Baseline | 402.41 (60.1780) | 419.21 (60.1780)
  PPT BL Change | 21.8583 (28.0167) | 4.3548 (28.0167)
Statistical Analysis 1: Comparison: rTMS and Exercise vs Sham rTMS and Exercise; PPT BL Change (treatment by time); Test type: Superiority; p = .6608, ANOVA — Threshold for statistical significance is P < .05; Repeated measures ANOVA with restricted maximum likelihood estimation and Kenward-Roger standard errors. DF = 45

5. Secondary Outcome: Timed Up & Go (TUG)
Description: Time in seconds to rise from a chair, walk 3 m, return and sit down
Time Frame: Within 1 hour post intervention
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | rTMS and Exercise | Sham rTMS and Exercise
Number analyzed (Participants) | 16 | 16
seconds
  TUG Baseline | 8.3919 (.4079) | 8.3056 (.4079)
  TUG BL Change | -.08021 (.803) | -.00542 (.1803)
Statistical Analysis 1: Comparison: rTMS and Exercise vs Sham rTMS and Exercise; Comparison of TUG BL Change (treatment by time); Test type: Superiority; p = .7706, ANOVA — Threshold for statistical significance is P < .05; Repeated measures ANOVA with restricted maximum likelihood estimation and Kenward-Roger standard errors. DF = 45

6. Secondary Outcome: Active Motor Threshold Motor Evoked Potential (AMT-MEP)
Description: The quadriceps active muscle responses (motor evoked potentials) that result from the single-pulse transcranial magnetic stimulation (TMS) pulses over the motor cortex. These AMT-MEP are measured peak-to-peak in microvolts (uV ). 10 AMT-MEP values were collected and averaged.
Time Frame: Within 1 hour post intervention
Population: 4 subjects withdrew from the study after the baseline measures. This left 16 subjects for the intervention arm of the study. A technical issue in how the TMS unit worked was discovered after collecting the first 4 subjects in the intervention part of the study. This impacted their AMT-MEP, ICF, and SICI data which were excluded from the analyses.
Measure: Least Squares Mean (Standard Error); unit: uV
Arm/Group | rTMS and Exercise | Sham rTMS and Exercise
Number analyzed (Participants) | 12 | 12
uV
  AMT-MEP Baseline | .1387 (.009634) | .1434 (.009634)
  AMT-MEP BL Change | -.00007 (.01107) | -.01441 (.01107)
Statistical Analysis 1: Comparison: rTMS and Exercise vs Sham rTMS and Exercise; Comparison of AMT-MEP BL Change (treatment by time); Test type: Superiority; p = .3665, ANOVA — Threshold for statistical significance is P < .05; Repeated measures ANOVA with restricted maximum likelihood estimation and Kenward-Roger standard errors. DF = 33

7. Secondary Outcome: Short Interval Cortical Inhibition (SICI)
Description: Transcranial magnetic stimulation (TMS), using the conditioning-test paired-pulse paradigm with a 3 ms interval, will be used. SICI is the ratio of the conditioning stimulus relative to the test stimulus. A ratio < 1.0 indicates inhibition.
Time Frame: Within 1 hour post intervention
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | rTMS and Exercise | Sham rTMS and Exercise
Number analyzed (Participants) | 12 | 12
ratio
  SICI Baseline | .5140 (.054) | .5996 (.1054)
  SICI BL Change | -.02588 (.07227) | -.1151 (.07227)
Statistical Analysis 1: Comparison: rTMS and Exercise vs Sham rTMS and Exercise; Comparison of SICI BL Change (treatment by time); Test type: Superiority; p = .3889, ANOVA — Threshold for statistical significance is P < .05; Repeated measures ANOVA with restricted maximum likelihood estimation and Kenward-Roger standard errors. DF = 33

8. Secondary Outcome: Intra Cortical Facilitation (ICF)
Description: Transcranial magnetic stimulation (TMS), using the conditioning-test paired-pulse paradigm with a 15 ms interval, will be used. ICF is the ratio of the conditioning stimulus relative to the test stimulus. A ratio > 1.0 indicates facilitation.
Time Frame: Within 1 hour post intervention
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | rTMS and Exercise | Sham rTMS and Exercise
Number analyzed (Participants) | 12 | 12
ratio
  ICF Baseline | 1.193 (.903) | .904 (.903)
  ICF BL Change | -.0354 (.1896) | .03042 (.1896)
Statistical Analysis 1: Comparison: rTMS and Exercise vs Sham rTMS and Exercise; Comparison of ICF BL Change (treatment by time); Test type: Superiority; p = .2192, ANOVA — Threshold for statistical significance is P < .05; Repeated measures ANOVA with restricted maximum likelihood estimation and Kenward-Roger standard errors. DF = 33

ADVERSE EVENTS:
Time Frame: From Baseline (Enrollment) until the end of Session 2, a total of approximately 3 weeks.
Arm/Group | rTMS and Exercise | Sham rTMS and Exercise
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT02881775/Prot_SAP_000.pdf